CLINICAL TRIAL: NCT03526848
Title: An Open Label, Randomized Study of the Safety and Antiretroviral Activity of 3BNC117 and 10-1074 in HIV-infected Individuals on Combination Antiretroviral Therapy and During Analytical Treatment Interruption.
Brief Title: 3BNC117 and 10-1074 in ART-treated Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Ragon Institute of MGH, MIT and Harvard (Other); Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCA-0965
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Human Immunodeficiency Virus
Keywords: 3BNC117; 10-1074; Broadly Neutralizing Antibody
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — 3BNC117 antibody; Antibodies, Monoclonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): HIV infected participants on ART will undergo analytical treatment interruption 2 days after the first infusion of 3BNC117 and 10-1074, and will receive 6 additional infusions of both antibodies at weeks 2, 4, 8, 12, 16 and 20 (Part A). Participants will remain off ART until week 38, if viral suppression is maintained (Part B).
  Interventions: Drug: 3BNC117; Drug: 10-1074; Other: Analytical treatment interruption
- Group 2 (Experimental): HIV infected participants on ART will remain on ART and will be administered seven infusions of 3BNC117 and 10-1074 at weeks 0, 2, 4, 8, 12, 16 and 20 (Part A). Analytical treatment interruption will begin at week 26 until week 38, if viral suppression is maintained (Part B).
  Interventions: Drug: 3BNC117; Drug: 10-1074; Other: Analytical treatment interruption

INTERVENTIONS:
Drug: 3BNC117 — Intravenous infusion of 3BNC117
  Other Names: Monoclonal antibody
Drug: 10-1074 — Intravenous infusion of 3BNC117
  Other Names: Monoclonal antibody
Other: Analytical treatment interruption — Analytical treatment interruption
  Other Names: ART interruption

SUMMARY:
The proposed study is a phase 1, open label, randomized study to evaluate the safety and antiretroviral activity of seven infusions of 3BNC117 and 10-1074, administered intravenously at 30 mg/kg dose level, in human immunodeficiency virus (HIV)-infected individuals on combination antiretroviral therapy (ART) and during an analytical interruption of ART.

DETAILED DESCRIPTION:
The proposed study is an open label study of the safety and antiretroviral activity of 3BNC117 and 10-1074 in HIV-infected individuals with well-controlled HIV infection on combination antiretroviral therapy (ART). 3BNC117 and 10-1074 are two broadly neutralizing antibodies (bNAbs) that target different sites on HIV-1 gp120. Our hypothesis is that the administration of repeated infusions of 3BNC117 and 10-1074 in the absence of ART will be safe and well tolerated, will maintain viral suppression in HIV-infected individuals during analytical treatment interruption (ATI) and will interfere with the maintenance of the HIV-1 reservoir.

Forty eligible participants will be randomized to either Group 1 or Group 2 in a 3:1 ratio:

Group 1 (n=30): participants will discontinue ART 2 days after the first infusion of 3BNC117 and 10-1074, and will receive 6 additional infusions of both antibodies at weeks 2, 4, 8, 12, 16 and 20 (Part A). Participants will remain off ART until week 38, if viral suppression is maintained (Part B).

Group 2 (n=10): participants will remain on ART and will be administered seven infusions of 3BNC117 and 10-1074 at weeks 0, 2, 4, 8, 12, 16 and 20 (Part A). ART will be discontinued at week 26 until week 38, if viral suppression is maintained (Part B).

After screening, participants will remain on ART and undergo leukapheresis, and will have the option to undergo LN biopsies 2-4 weeks prior to first 3BNC117 and 10-1074 infusions.

Participants enrolled in group 1 will discontinue their ART 2 days after the first 3BNC117 and 10-1074 infusions. Participants enrolled in group 2 will discontinue their ART at week 26. If the participant's ART regimen includes an NNRTI, the NNRTI will be switched to an integrase inhibitor-based regimen, 4 weeks prior discontinuing all antiretroviral drugs.

During the ATI periods of the study, ART will be resumed if there is a > 30% decline in CD4+ T cell count or CD4+ T cell count decreases to < 350 cells/μl from baseline (day 0) and these changes are confirmed during next visit. ART will also be re-initiated if the participant develops symptoms of severe acute retroviral syndrome or becomes pregnant. In addition, ART will be resumed according the following virologic parameters:

Part A (wk 0 - wk 26), ART will be resumed if group 1 participants have 2 consecutive plasma HIV-1 RNA levels > 200 copies/ml.

Part B (wk 26 - wk 38), ART will be resumed if group 1 or group 2 participants have sustained (> 4 weeks) HIV-1 RNA levels > 1,000 copies/ml.

Part C (wk 38 - wk 48), group 1 and group 2 participants who have not met criteria to reinitiate ART will be offered to continue off ART with close monitoring. In Part C, ART will be resumed if the participant has 2 consecutive plasma HIV-1 RNA levels > 1,000 copies/ml.

All participants will be followed for a total of 48 weeks from enrollment (day 0). Participants will be invited to return for a large blood draw after they reach at least 24 weeks of viral suppression after ART is re-initiated, if this occurs after the active study follow up period.

Safety assessments will be performed at multiple time points following 3BNC117 and 10-1074 infusions. The effects of 3BNC117 and 10-1074 infusions on the HIV-1 reservoir of ART-suppressed HIV-infected individuals will be evaluated by several assays. These evaluations will occur at baseline (day 0) and at week 26.

ELIGIBILITY:
Inclusion Criteria:

* Male and females, age 18 to 65.
* Confirmed HIV-1 infection.
* On antiretroviral therapy with plasma HIV-1 RNA levels of < 50 copies/ml for at least 12 months, and < 20 copies/ml at screening. Note: a single viral load measurement > 50 but < 500 copies/ml during this time period is allowed.
* Current CD4+ T cell counts > 500 cells/μl and CD4+ T cell count nadir of > 200 cells/μl.
* If on an NNRTI-based regimen, willing to switch to an integrase inhibitor-based regimen for at least 4 weeks prior to discontinuing ART
* If sexually active male or female, participating in sexual activity that could lead to pregnancy and of reproductive potential, agrees to follow the contraception requirements outlined Section 6.12.12 Family Planning Counseling. Participants should also agree to use a male or female condom while off ART to prevent infecting sexual partners.

Exclusion Criteria:

* Have a history of AIDS-defining illness within 3 years prior to enrollment.
* History of systemic corticosteroids (long term use), immunosuppressive anti-cancer, interleukins, systemic interferons, systemic chemotherapy or other medications considered significant by the trial physician within the last 6 months.
* Any clinically significant acute or chronic medical condition (such as autoimmune diseases), other than HIV infection, that in the opinion of the investigator would preclude participation.
* Hepatitis B or C infection as indicated by the presence of Hepatitis B surface antigen (HBsAg) or hepatitis C virus RNA (HCV-RNA) in blood.
* History of resistance to 2 or more classes of antiretroviral medication.
* Laboratory abnormalities in the parameters listed below:
* Absolute neutrophil count ≤ 1,000 cells/μl
* Hemoglobin ≤ 10 gm/dL
* Platelet count ≤ 100,000 cells/μl
* Alanine aminotransferase (ALT) ≥ 1.5 x ULN
* Aspartate aminotransferase (AST) ≥ 1.5 x ULN
* Alkaline phosphatase ≥ 1.5 x ULN
* Total bilirubin ≥ 1.5 x ULN
* eGFR < 60 mL/min/1.73m2
* Prothrombin time (PT) > 1.2 x upper limit of normal (ULN). (only if LN biopsies are performed)
* Partial Thromboplastin Time (PTT) > 1.2 x upper limit of normal (ULN) (only if LN biopsies are performed)
* Pregnancy or lactation
* Receipt of any therapeutic HIV vaccine or anti-HIV monoclonal antibody therapy in the past.
* Participants with known hypersensitivity to any constituent of the investigational products.
* Participation in another clinical study of an investigational product currently or within past 12 weeks, or expected participation during this study.
* History of intolerance, sensitivity, allergy or anaphylaxis to benzodiazepines or other narcotics to be used during LN biopsy. (only if LN biopsies are performed)
* Previous adverse reaction or allergy to lidocaine or other amide anesthetics, as well as benzocaine or other ester type anesthetics. (only if LN biopsies are performed)
* History of underlying medical condition for which antibiotic prophylaxis for invasive procedures is required (only if LN biopsies are performed)
* Currently taking anticoagulants including but not limited to: heparin (Hep-Lock, Hep-Pak, Hep-Pak CVC, Heparin Lock Flush), warfarin (Coumadin), tinzaparin (Innohep), enoxaparin (Lovenox), danaparoid (Orgaran), dalteparin (Fragmin), clopidogrel (Plavix), dipyridamole (Persantine), fondaparinux (Arixtra), argatroban (Agratroban), and bivalrudin (Angiomax). Prophylactic aspirin and regular NSAID use permitted. (only if LN biopsies are performed)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
The change in the size of the functional, latent HIV-1 reservoir between baseline and after seven infusions of 3BNC117 and 10-1074 | Day 0 and week 26
  The size of the functional, latent HIV-1 reservoir is determined by the number of infectious units per 106 resting memory CD4+ T cells (IUPM) using a viral outgrowth assay at baseline and after seven infusions of 3BNC117 and 10-1074
The size of the proviral HIV-1 reservoir | 48 weeks
  Size of the proviral HIV-1 reservoir as determined by total HIV-1 DNA and integrated HIV-1 DNA in circulating total CD4+ T cells before and after seven infusions of 3BNC117 and 10-1074.
The rate of viral rebound | Week 12 (group 1) and week 38 (group 2)
  Rate of viral rebound (plasma HIV-1 RNA level > 200 copies/ml in 2 consecutive measurements) or indication to reinitiate ART at 12 weeks after ART interruption (study week 12 in group 1, study week 38 in group 2).
Time to return of HIV-1 viremia | 48 weeks
  Time to return of HIV-1 viremia (plasma HIV-1 RNA level > 200 copies/ml in 2 consecutive measurements) after ART interruption.
The rate of adverse events (AE) and serious adverse events (SAE). | 48 weeks
  The rate of adverse events (AE) and serious adverse events (SAE).
The severity of adverse events (AE) and serious adverse events (SAE). | 48 weeks
  The severity of adverse events (AE) and serious adverse events (SAE).

SECONDARY OUTCOMES:
The rate of viral rebound at 26 weeks after ART interruption in group 1. | 26 weeks
  Rate of viral rebound (plasma HIV-1 RNA level > 200 copies/ml in 2 consecutive measurements) at 26 weeks after ART interruption in group 1.
Serum levels of 3BNC117 and 10-1074 at the time of viral rebound | 48 weeks
  Serum levels of 3BNC117 and 10-1074 at the time of viral rebound

CONTACTS AND LOCATIONS:
Overall Officials: Marina Caskey, MD, Study Chair — The Rockefeller University
Locations (2):
- United States (2):
  - Ragon Institute of MGH, MIT, and Harvard, Boston, Massachusetts
  - The Rockefeller University, New York, New York

IPD SHARING:
Plan to Share IPD: No